CLINICAL TRIAL: NCT05805436
Title: The Use of Preoperative Osmotic Laxatives to Improve Recovery of Bowel Function After Robotic-assisted Urologic Surgery
Brief Title: Preop Laxatives in Robotic Urologic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chad R. Tracy (Other)
Responsible Party: Sponsor-Investigator, Chad R. Tracy, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202209015
Record Dates: First submitted 2023-03-03; First posted 2023-04-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Kidney Cancer; Constipation
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Constipation | interventions — polyethylene glycol 3350

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Do not receive polyethylene glycol before surgery
- Intervention (Experimental): Receive polyethylene glycol before surgery
  Interventions: Drug: Polyethylene Glycol 3350

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — Patients in the intervention arm will take polyethylene glycol 3350 for three days before robotic urologic surgery. Patients in the control arm will not.
  Arms: Intervention

SUMMARY:
Minimally-invasive surgery, either laparoscopic or robotic, is commonly used in urology. Several urologic procedures including prostatectomy, radical nephrectomy, and partial nephrectomy are now commonly performed robotically. Patients undergoing these procedures often have delayed return of bowel function and persistent gastrointestinal symptoms including nausea/vomiting, abdominal distension, and bloating for several days to weeks after surgery. Postoperative stool softeners and laxatives are routinely used in an effort to minimize these symptoms, with varying degrees of success. The aim of this study will be to evaluate whether the use of a preoperative osmotic laxative will be beneficial in improving recovery of bowel function and alleviating postoperative gastrointestinal complaints in patients undergoing these procedures. Patients will be randomized to either receive or not receive three days of polyethylene glycol (PEG, also known as MiraLAX) on the three days before surgery. Patients in both groups will receive the same postoperative bowel regimen including scheduled PEG both in the hospital and upon discharge until first bowel movement. Patients will be given a questionnaire and diary to record their postoperative gastrointestinal symptoms and time to first bowel movement. These questionnaires and diaries will then be analyzed to determine differences in time to first bowel movement and gastrointestinal complaints during their recovery from surgery.

ELIGIBILITY:
Inclusion criteria:

-Patients 30 years or older undergoing robotic-assisted laparoscopic radical prostatectomy, transperitoneal radical nephrectomy, or transperitoneal partial nephrectomy

Exclusion criteria:

* Patients under 30 years old
* Patients with a contraindication to receiving polyethylene glycol or other forms of laxatives
* People who regularly take Miralax
* Patients undergoing retroperitoneal radical or partial nephrectomy
* Patients with severe ulcerative colitis or Crohn's disease
* Patients with intestinal diversions (colostomy, ileostomy)
* Patients with prior abdominal or pelvic radiation
* Patients who will not follow up with UIHC postoperatively
* Patients who are incarcerated

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Time to first bowel movement after surgery | 7 days
  Time to first bowel movement after surgery

SECONDARY OUTCOMES:
Narcotic usage | 7 days
  Morphine equivalents used by patients in the first 7 days postoperatively
Patient Assessment of Constipation-Symptoms (PAC-SYM) Questionnaire | 7 days
  Patient Assessment of Constipation-Symptoms (PAC-SYM) Questionnaire scores 7 days postoperatively (scale 0 - 48, higher score indicates worse constipation)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States